CLINICAL TRIAL: NCT05020535
Title: Biomarker and Edema Attenuation in IntraCerebral Hemorrhage (BEACH) Phase 2a Trial
Brief Title: Biomarker and Edema Attenuation in IntraCerebral Hemorrhage (BEACH)
Acronym: BEACH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: University of Kentucky (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00295926; 1R01AG069930-01 (NIH); R01AG069930 (NIH)
Record Dates: First submitted 2021-08-19; First posted 2021-08-25 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Intracerebral Hemorrhage
Keywords: Intracerebral hemorrhage; MW01-6-189WH; MW189; Radiographic perihematomal edema; Neuroinflammation; Cerebral edema
MeSH Terms: conditions — Cerebral Hemorrhage; Neuroinflammatory Diseases; Brain Edema | interventions — TT-301; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Parallel 1:1
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, study staff, analytic staff (to patient identifiers), sponsor staff (only to treatment allocation, unblinded to enable handling and review of data and drug accountability prior to database lock)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): MW189 (0.25 mg/kg) is administered within 24 hours of symptom onset and every 12 hours for up to 5 days (10 total doses) or until discharge (if earlier than 5 days)
  Interventions: Drug: MW189
- Control (Placebo Comparator): Administration of saline within 24 hours of symptom onset and every 12 hours for up to 5 days (10 total doses) or until discharge (if earlier than 5 days)
  Interventions: Other: Saline

INTERVENTIONS:
Drug: MW189 — MW189 (0.25 mg/kg) is administered within 24 hours of symptom onset and every 12 hours for up to 5 days (10 total doses) or until discharge (if earlier than 5 days)
  Arms: Experimental
Other: Saline — Administration of saline within 24 hours of symptom onset and every 12 hours for up to 5 days (10 total doses) or until discharge (if earlier than 5 days)
  Arms: Control

SUMMARY:
This first-in-patient phase 2a pilot study will assess the safety and tolerability of MW01-6-189WH (hereafter called MW189) in patients with Intracerebral Hemorrhage (ICH).

DETAILED DESCRIPTION:
This first-in-patient phase 2a pilot study will assess the safety and tolerability of MW01-6-189WH (hereafter called MW189) in patients with Intracerebral Hemorrhage (ICH).

This study will monitor exploratory radiographic and clinical endpoints, explore the use of biochemical biomarkers to demonstrate target engagement and biological response to a potential new therapy targeted to neuroinflammation and synaptic dysfunction mechanisms.

MW189 is a novel small molecule drug candidate developed as a selective suppressor of disease-and injury-induced proinflammatory cytokine overproduction associated with destructive neuroinflammation/synaptic dysfunction cycles. In animal models of acute brain injuries such as ICH and Traumatic Brain Injury (TBI), MW189 attenuates neuroinflammation, reduces cerebral edema, and improves functional and cognitive performance. The investigators seek to establish if these targets are modified in humans with ICH.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of spontaneous, non-traumatic ICH.
* 10 mL ≤ ICH ≤ 60 mL (confirmed via diagnostic and stability CT scans utilizing volumetric assessment)
* Participants receiving anticoagulants are eligible upon reversal and stability within 24hrs after onset of ICH symptoms
* Age ≥ 18 years
* Able to receive first dose of test article ≤ 24h after onset of ICH symptoms
* NIHSS score ≥ 2 at randomization or Glasgow Coma Scale ≥ 5 at randomization
* Controlled blood pressure (systolic BP < 180 mm Hg) at randomization.
* Premorbid magnetic resonance spectroscopy (mRS) of 0-2
* Has adequate venous access
* No planned surgical intervention except EVD
* Written informed consent from the patient or legally authorized representative (LAR)

Exclusion Criteria:

* Unstable hematoma defined as > 6 mL increase as compared to previous CT volume taken at least 6 hours apart within 24 hrs after onset of ICH symptoms.
* Anticipated neurosurgical evacuation by open surgery or minimally invasive surgery with or without Alteplase (EVD allowed).
* Uncontrolled temp >38.5˚C at enrollment.
* Signs of intracranial infection or emergence of a systemic infection
* Is pregnant or lactating
* Signs of liver and kidney chronic disease (i.e. creatinine >2, bilirubin > 3, receiving dialysis)
* Non-reversible bleeding diathesis
* Used any chronic immunosuppressants or chronic anti-inflammatory drugs (excluding low-dose aspirin), by any route of administration within the past 7 days.
* Anticipated withdrawal of life-sustaining therapies within the first week after admission.
* In the opinion of the investigator, patient has any contraindication to the planned study assessments.
* In the opinion of the investigator, patient has a condition that could interfere with the proposed treatment or unacceptably increase the individual's risk by participating in the study.
* Concomitant enrollment in another acute interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Difference in the proportion of all cause-morality between arms | 7 days post-randomization
  Assess the safety and tolerability of MW189 for patients as determined by the rate of death during the treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Van Eldik, Principal Investigator — University of Kentucky
Locations (11):
- United States (11):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Stanford University, Palo Alto, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - Cleveland Clinic Florida, Stuart, Florida
  - University of Kentucky, Lexington, Kentucky
  - Johns Hopkins Hospital, Baltimore, Maryland
  - University of New Mexico, Albuquerque, New Mexico
  - New York University Grossman School of Medicine, Brooklyn, New York
  - University of Cincinnati, Cincinnati, Ohio
  - University of Texas Houston, Houston, Texas
  - University of Texas San Antonio, San Antonio, Texas

REFERENCES:
- [Derived] Sorensen G, Remillard W, Schlechter M, Kampp M, Whisler Brady C, Kildahl K, Mould A, Ziai W, Lane K, Van Eldik LJ, Distasio A, Lu J, Sansing LH, Hanley DF, Magid-Bernstein J. Operationalizing a complex acute clinical trial: Lessons from the BEACH study. J Clin Transl Sci. 2025 Sep 12;9(1):e215. doi: 10.1017/cts.2025.10152. eCollection 2025. PMID 41040632
- [Derived] Sorensen G, Remillard W, Schlechter M, Kampp M, Sansing LH, Brady CW, Kidahl K, Ziai W, Van Eldik L, Distasio A, Lu J, Magid-Bernstein J, Hanley D. Operationalizing a complex acute clinical trial: Lessons from the BEACH study. medRxiv [Preprint]. 2025 Mar 31:2025.03.28.25324776. doi: 10.1101/2025.03.28.25324776. PMID 40236420